CLINICAL TRIAL: NCT03749655
Title: A Feasibility Study Assessing the Inclusion of Physical Activity Promotion to Standard Care Pulmonary Rehabilitation and Cognitive Behavioural Therapy in Patients With COPD Who Are Anxious and Depressed
Brief Title: Physical Activity Promotion Added to Standard Care Pulmonary Rehabilitation and Cognitive Behavioural Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08968
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Rehabilitation; Physical activity; Anxiety and depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Single centre feasibility, single blind, parallel, randomised controlled study.
Masking Description: Principle investigator will be blinded from the randomisation as this member will conduct CBT with all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR+CBT (No Intervention): Standard care Pulmonary rehabilitation will be given alongside cognitive behavioural therapy
- PR+CBT+PA Promotion. (Experimental): Standard care Pulmonary rehabilitation will be given alongside cognitive behavioural therapy and physical activity promotion.
  Interventions: Behavioral: Physical Activity Promotion

INTERVENTIONS:
Behavioral: Physical Activity Promotion — The physical activity (PA) promotion intervention will be provided only to the intervention group, and will include: 1) a step-counter with a digital display, 2) an interview discussing motivational issues, favourite daily activities and strategies to become more physically active; and 3) a tailored physical activity coaching plan including an Individualised activity goal (in steps/day) revised twice weekly through consultation sessions (16 sessions in total). Patients' targets will be revised twice weekly during the consultation sessions which will be incorporated into the Pulmonary rehabilitation sessions. The aim is to increase physical activity by 10% each week. The goal can be altered if required.
  Arms: PR+CBT+PA Promotion.

SUMMARY:
In patients with Chronic Obstructive Pulmonary Disease (COPD) daily physical activity is reduced compared to healthy age-matched individuals. Reduced levels of physical activity in patients with COPD are associated with increased risk for exacerbations, hospital admissions and mortality.

Pulmonary rehabilitation (PR) constitutes standard care for patients with COPD as it improves exercise capacity, quality of life and reduces the risk for exacerbation and hospitalisation. Participation in PR, however, does not necessarily translate into improved daily physical activity levels. It is currently uncertain whether addition of physical activity promotion strategies to standard PR programs induces an improvement in daily physical activity along with exercise capacity and quality of life compared to pulmonary rehabilitation alone.

Physical activity (PA) is a complex health behaviour that is modified by behavioural change interventions. PA promotion programs through the use of wearable monitors (i.e. pedometers, accelerometers) with goal setting and feedback, have shown to increase daily physical activity, but not exercise capacity or quality of life in COPD patients. Therefore, combination of both PR and PA promotion strategies is necessary to translate PR-induced improvements in functional capacity into improved daily physical activity level. The investigators propose to perform a feasibility study assessing patient adherence to PA promotion incorporated into a standard PR program. To enhance adherence to the PA promotion strategy, Cognitive Behavioural Modification Strategies (CBM) will be provided to patients undertaking PR. CBM strategies facilitate the goals of PR as they address several behavioural barriers including anxiety, depression and physical inactivity, and constitutes an important component in the management of COPD to improve engagement with PR and promote a physically active lifestyle. The investigators will divide patients into two programs: one including PR, PA promotion and CBM and the other comprising standard PR and CBM provision. The investigators will compare patients' adherence (16 sessions of PR) to both programs.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a debilitating and progressive disease, primarily affecting the respiratory system. In many patients, it also has adverse extra-pulmonary effects, such as skeletal muscle dysfunction and weakness (Maltais, et al. 2014). Pulmonary and skeletal muscle metabolic abnormalities enhance the ventilatory requirement during exercise, resulting in exercise-associated symptoms such as breathlessness and leg discomfort. These symptoms make every day physical activity an unpleasant experience, which many patients try to avoid (Troosters, et al. 2013). Physical activity levels are therefore remarkably lower in COPD patients than healthy age-matched individuals, presenting a major predictor of exacerbations, hospitalisations and mortality and in these patients (Pitta et al. 2005) & (Garcia-Aymerich et al. 2006).

Implementation of exercise training as part of Pulmonary Rehabilitation aims to reverse the systemic consequences of COPD, in particular skeletal muscle dysfunction and weakness (Troosters, et al. 2013) . Currently pulmonary rehabilitation programs have shown substantial improvements in exercise capacity; however, these findings have not consistently progressed into improvements in daily levels of physical activity (Watz et al. 2014). One reason for this may link to physical activity in COPD being a complex health behaviour (Troosters, et al. 2013).

Recently, physical activity coaching, including weekly targets and feedback, has shown to be effective in patients with COPD in terms of improving daily steps over a period of three months (Lahham et al. 2016). Accordingly, activity coaching may be added to standard pulmonary rehabilitation to facilitate the rehabilitation-induced improvements in exercise capacity to progress into improvements in physical activity (Lahham et al. 2016).

Alongside the physical barriers influencing daily physical activity, the distressing nature of COPD has a significant impact on patients' psychological well-being. Major focusing points for COPD patients are the sense of feeling unwell, the inability to perform everyday activities and the emotional consequences of the condition. These symptoms can promote anxiety and depression, which are prevalent in patients with COPD, are associated with poorer treatment outcomes, and reduced survival (Ng, T-P et al. 2007).

Cognitive Behavioural Modification (CBM) strategies constitute an intervention that focuses on understanding how experiences are interpreted. It provides an understanding of the interaction between thoughts, mood, behaviour and physical sensations, which are intrinsically linked [8]. Techniques used for anxiety include education on anxiety and COPD, planning/pacing, distraction techniques, breathing control, relaxation and managing worry. These techniques help to break the vicious cycle of anxiety and can reduce patients' distress (Heslop & Foley. 2009).

Similar techniques for patients suffering mainly from depression include education about depression and physical inactivity and planning and recording activities each day, while rating these for achievement or pleasure. These techniques help to break patient inactivity, which can lead to low mood and poor physical condition. A key treatment for depression can involve encouragement to increase activities within the patients' physical capabilities. A study found clinical and statistically significant improvements in anxiety and depression scores and a statistically significant reduction in hospital admissions following CBM. CBM is therefore an important approach to incorporate into COPD management to improve engagement with both pulmonary rehabilitation and the physical activity promotion programme Heslop & Foley. 2009.

The efficacy of incorporating a physical activity promotion program to standard care pulmonary rehabilitation along with CBM strategies is still unknown. Accordingly, it is proposed to study patient compliance with the physical activity promotion programme comprising weekly goals in terms of daily step counts measured by a commercially available step counter. Compliance to the intervention is defined as at least 4 days per week (> 8 hours/day) with valid step count data (>70 steps/day) ensuring that patients use the step counter on a daily basis. Over the 8-week program patients should have a minimum of 6 weeks (75%) compliance with the physical activity intervention. If patients adhere adequately to this programme, a randomised controlled trial will be designed to study the long-term effects of adding physical activity promotion to Pulmonary Rehabilitation (including exercise training, education, physical activity promotion and behavioural modification strategies) on the risk for COPD exacerbations and hospitalisations.

ELIGIBILITY:
Inclusion Criteria:

* COPD confirmed by obstructive spirometry
* Clinically stable male or female COPD patients aged 40 years or older
* Optimised medical therapy
* Able to provide informed consent
* HADS score of 8 and above

Exclusion Criteria:

* Orthopaedic, neurological or other concomitant diseases that significantly impair normal biomechanical movement patterns, as judged by the investigator.
* Moderate or severe COPD exacerbation (AECOPD) within 4 weeks.
* Unstable ischaemic heart disease, including myocardial infarction within 6 weeks.
* Moderate or severe aortic stenosis or hypertrophic obstructive cardiomyopathy.
* Uncontrolled hypertension.
* Another condition likely to limit life expectancy to less than one year (principally metastatic malignancy).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Patient compliance with the physical activity promotion intervention | 8 weeks (16 sessions)
  Whether patients use the step counter for an 8 week period of physical activity promotion while undertaking pulmonary rehabilitation. Compliance to the intervention is defined as at least 4 days per week with valid step count data (>70 steps/day). Over the 8-week program patients should have a minimum of 6 weeks (75%) compliance with the physical activity intervention.
Patient Experience of Physical Activity | Measured 1 week prior and 1 week post rehabilitation
  Measured using the innovative Clinical Visit of COPD Questionnaire (C-PPAC)

SECONDARY OUTCOMES:
Change in daily physical activity. | Measured 1 week prior and 1 week post rehabilitation
  Measured via steps/day using a triaxial accelerometer
Change in symptoms of anxiety and depression. | Measured 1 week prior and 1 week post rehabilitation
  Assessed using the Hospital Anxiety and Depression Scale (HADS) questionnaire. Scale measures for Anxiety and Depression are both out of 21. Scoring is grouped as: Normal= 0-7, Borderline abnormal= 8-10, 11-21= Abnormal.
  For the investigators study a score for Anxiety and/or depression of >8 is required at inclusion.
Change in functional capacity | Measured 1 week prior and 1 week post rehabilitation
  Assessed by the 6-min walk test
Change in quality of life | Measured 1 week prior and 1 week post rehabilitation
  Assessed using COPD Assessment Test (COPD)
Change in quality of life | Measured 1 week prior and 1 week post rehabilitation
  Assessed using the clinical COPD questionnaire (CCQ). The total CCQ score is calculated by adding the scores of the ten items and dividing that number by 10. The scale varies between 0 (very good health) to 6 (extremely poor health status).

CONTACTS AND LOCATIONS:
Locations (1):
- Newcastle upon Tyne NHS trust, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Troosters T, van der Molen T, Polkey M, Rabinovich RA, Vogiatzis I, Weisman I, Kulich K. Improving physical activity in COPD: towards a new paradigm. Respir Res. 2013 Oct 30;14(1):115. doi: 10.1186/1465-9921-14-115. PMID 24229341
- [Background] Pitta F, Troosters T, Spruit MA, Probst VS, Decramer M, Gosselink R. Characteristics of physical activities in daily life in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 May 1;171(9):972-7. doi: 10.1164/rccm.200407-855OC. Epub 2005 Jan 21. PMID 15665324
- [Background] Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM. Regular physical activity reduces hospital admission and mortality in chronic obstructive pulmonary disease: a population based cohort study. Thorax. 2006 Sep;61(9):772-8. doi: 10.1136/thx.2006.060145. Epub 2006 May 31. PMID 16738033
- [Background] Watz H, Pitta F, Rochester CL, Garcia-Aymerich J, ZuWallack R, Troosters T, Vaes AW, Puhan MA, Jehn M, Polkey MI, Vogiatzis I, Clini EM, Toth M, Gimeno-Santos E, Waschki B, Esteban C, Hayot M, Casaburi R, Porszasz J, McAuley E, Singh SJ, Langer D, Wouters EF, Magnussen H, Spruit MA. An official European Respiratory Society statement on physical activity in COPD. Eur Respir J. 2014 Dec;44(6):1521-37. doi: 10.1183/09031936.00046814. Epub 2014 Oct 30. PMID 25359358
- [Background] Lahham A, McDonald CF, Holland AE. Exercise training alone or with the addition of activity counseling improves physical activity levels in COPD: a systematic review and meta-analysis of randomized controlled trials. Int J Chron Obstruct Pulmon Dis. 2016 Dec 8;11:3121-3136. doi: 10.2147/COPD.S121263. eCollection 2016. PMID 27994451
- [Background] Ng TP, Niti M, Tan WC, Cao Z, Ong KC, Eng P. Depressive symptoms and chronic obstructive pulmonary disease: effect on mortality, hospital readmission, symptom burden, functional status, and quality of life. Arch Intern Med. 2007 Jan 8;167(1):60-7. doi: 10.1001/archinte.167.1.60. PMID 17210879
- [Background] Heslop K, Foley T. Using cognitive behavioural therapy to address the psychological needs of patients with COPD. Nurs Times. 2009 Sep 29-Oct 5;105(38):18-9. PMID 19860064
- [Derived] Armstrong M, Hume E, McNeillie L, Chambers F, Wakenshaw L, Burns G, Marshall KH, Vogiatzis I. Behavioural modification interventions alongside pulmonary rehabilitation improve COPD patients' experiences of physical activity. Respir Med. 2021 Apr-May;180:106353. doi: 10.1016/j.rmed.2021.106353. Epub 2021 Mar 9. PMID 33735798

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT03749655/Prot_ICF_000.pdf